CLINICAL TRIAL: NCT07352358
Title: Randomized Trial of Anticoagulation Plus Batroxobin for Acute Cerebral Venous Thrombosis (ABACVT)
Brief Title: Randomized Trial of Anticoagulation Plus Batroxobin for Acute Cerebral Venous Thrombosis
Acronym: ABACVT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Meng Ran, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMeng3
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Venous Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Batroxobin; Anticoagulants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- batroxobin plus anticoagulation (Experimental): The experimental group adopted the combined use of anticoagulants (low molecular weight heparin bridged to warfarin 3 mg/day, rivaroxaban 10-20 mg/day or dabigatran 110-150 mg twice daily) and batroxobin (initial dose of 10 BU, followed by 5 BU every other day).
  Interventions: Drug: batroxobin; Drug: Anticoagulation Agents
- standard anticoagulation treatment group (Active Comparator): Use anticoagulants (bridge with low-molecular-weight heparin to warfarin 3 mg/day, rivaroxaban 10-20 mg/day or dabigatran 110-150 mg twice daily)
  Interventions: Drug: Anticoagulation Agents

INTERVENTIONS:
Drug: batroxobin — The initial dose of batroxobin is 10 BU, followed by 5 BU every other day.
  Arms: batroxobin plus anticoagulation
Drug: Anticoagulation Agents — Low-molecular-weight heparin bridging to warfarin 3 mg/day, rivaroxaban 10-20 mg/day or dabigatran 110-150 mg twice daily.

SUMMARY:
A total of 72 patients meeting the diagnostic criteria for acute cerebral venous thrombosis were included in this study. A multi-center stratified randomization method was adopted, with the stratification factor being each participating center. There were three groups in total, and within each group, the experimental group and the control group were assigned in a 1:1 ratio. Finally, all the experimental groups and control groups were combined to form the overall experimental group and control group. Random sequences were generated using a computer random number generator, and concealed allocation was implemented using sealed, opaque, consecutively numbered envelopes. Patients and their families, researchers, treating physicians and nurses, outcome assessors, and other personnel directly involved in the trial were unaware of the treatment allocation. Patients meeting the inclusion criteria for acute CVT were immediately given standard anticoagulant therapy (subcutaneous injection of low-molecular-weight heparin at a dose of 0.4 mg every 12 hours for 5-7 days). Subsequently, patients were randomly assigned to the experimental group and the control group. The experimental group received a combination of anticoagulants (low-molecular-weight heparin bridged to warfarin 3 mg/day, rivaroxaban 10-20 mg/day, or dabigatran 110-150 mg twice daily) and batroxobin (initial dose of 10 BU, followed by 5 BU every other day); the control group received only the aforementioned anticoagulants. Follow-up evaluations were conducted at 7 days, 30 days, and 90 days after baseline. Baseline data included demographic characteristics, routine laboratory tests (complete blood count, liver and kidney function tests, electrolyte analysis, urine analysis, and coagulation function), TOF MRV, NIHSS score, and mRS score. Follow-up data covered TOF MRV, NIHSS score, and mRS score at 7 days, 30 ± 7 days, and 90 ± 7 days for the treatment groups. NIHSS and mRS assessments were conducted by neurologists who were unaware of the treatment plan. To minimize potential bias in the primary outcome, qualified personnel at each research center reviewed the 90-day clinical evaluations according to a standardized procedure manual. To ensure the validity and reproducibility of the evaluations, training courses were held for all researchers at each center. In addition, researchers recorded in detail the concomitant medications and adverse events that occurred within 90 days after patient enrollment. The primary endpoint was the proportion of patients achieving recanalization within 7 days of treatment. Secondary endpoints included the proportion of patients achieving neurological improvement (NIHSS score reduction ≥ 2 points) or deterioration (NIHSS score increase ≥ 4 points) at 7 days, 30 days, and 90 days, the proportion of patients achieving functional improvement (mRS score reduction) within 90 days, and the occurrence of CVT recurrence or other vascular events within 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Neuroimaging confirmed acute CVT;
3. Symptoms onset was within 30 days prior to enrollment;
4. Signed the informed consent form.

Exclusion Criteria:

1. Patients with bleeding (including those with bleeding disorders due to coagulation and vascular disorders, active peptic ulcers, suspected intracranial hemorrhage, thrombocytopenic purpura, hemophilia, during menstruation, during surgery, urinary tract bleeding, hemoptysis, premature delivery, miscarriage, women immediately after delivery and during the puerperium with bleeding from the sexual organs, etc.);
2. Recently operated patients
3. Patients with a potential for bleeding (such as those with visceral tumors, diverticulitis of the digestive tract, colitis, subacute bacterial endocarditis, severe hypertension, and severe diabetes, etc.);
4. Those who are currently taking anticoagulant drugs and platelet function inhibitors (such as aspirin) and those who are using antifibrinolytic agents;
5. Those with a pre-medication fibrinogen concentration lower than 100 mg/dl;
6. Patients with severe liver or kidney dysfunction and other conditions such as papillary muscle rupture, ventricular septal perforation, cardiogenic shock, and multiple organ failure.
7. Those who have a history of allergy to this preparation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving complete recanalization at day 7 | On the seventh day after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No